CLINICAL TRIAL: NCT00466349
Title: International Spinal Muscular Atrophy Patient Registry
Brief Title: International SMA Patient Registry
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Cure SMA (Other)
Responsible Party: Principal Investigator, Tatiana Foroud, Department Chair, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 0202-03
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Muscular Atrophy, Spinal
Keywords: SMA Type I; SMA Type II; SMA Type III; SMN; Werdnig-Hoffman Disease; Spinal Muscular Atrophy; Registry; SMA Type IV
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a registry of individuals affected by Spinal Muscular Atrophy (SMA) and/or family members of individuals affected by SMA. The purpose of the registry is to allow researchers studying the biological basis of SMA and potential therapies in SMA access to individuals interested in participating in research and/or experimental therapies. The International SMA Patient Registry is supported by CureSMA.

DETAILED DESCRIPTION:
This project is supported by CureSMA (http://curesma.org/).

The Registry functions as a liaison between patients and families interested in participating in research and researchers interested in studying SMA. The Registry contains information from 2,500 families and over 3,000 individuals with SMA from all over the world and continues to grow.

The Registry has helped recruit participants for clinical trials and has provided data for important SMA research studies. The Registry helps centralize information on this rare genetic disease, provides families a way to learn about research studies and provides researchers a way to find research participants.

Individuals and families affected by SMA are invited to join the Registry. Participants are asked to complete questionnaires about the symptoms, treatment, medications, and other experiences with SMA. Visit the Participant Portal for more information on how to sign up for the Registry.

Participant information is stored in a secure database. Researchers who are interested in studying SMA can request two types of data from the Registry, de-identified information and identifiable information. De-identified information does not contain any names or personal identifiers, and can be given to researchers without having to contact Registry families. Identifiable information includes information that can identify you and will never be released without getting your written permission to do so. Identifiable information includes data such as names and dates of birth. Some researchers may also request contact with families to obtain specific information or to request participation in a research study. In these instances, the Registry will contact each potential participant to ask if they are willing to share their identifiable information for a research project.

The Registry recognizes the importance of global collaboration. Working together with researchers from all over the world is very important in the investigation of SMA. In 2008 the Registry joined the group, Translational Research in Europe for the Assessment and Treatment of Neuromuscular Diseases (TREAT-NMD) in a global collaboration to further the research goals of the neuromuscular disease community. TREAT-NMD has developed a global database that compiles deidentified data transferred from participating registries around the world. The main objective of the TREAT-NMD database is to assess the feasibility of clinical trials, to facilitate the planning of clinical trials and to support the enrollment of patients in clinical trials. This international database will also be used to answer questions regarding the prevalence of particular neuromuscular disorders and assessing the support of other activities such as assessing standards of care and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals or family members of individuals who have been diagnosed with SMA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals or family members of individuals who have been diagnosed with SMA.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 1986-05; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Study is a patient registry | unlimited

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Foroud, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States